CLINICAL TRIAL: NCT05403983
Title: MOM-mi: Exploring the Effectiveness of a 12-week Movement Intervention on Heart Rate Variability and Self-compassion Among New Mothers
Brief Title: Effectiveness of a 12-week Movement Intervention on Heart Rate Variability and Self-compassion Among New Mothers
Acronym: MOM-mi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Fraser Valley (Other)
Collaborators: Les Mills International (Unknown)
Responsible Party: Principal Investigator, Gillian Hatfield, Associate Professor, University of the Fraser Valley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101075
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In person movement intervention (Experimental): In person yoga movement intervention (Les Mills BodyBalance: mixture of yoga, tai chi, pilates) two times per week
  Interventions: Behavioral: Yoga movement intervention
- Online yoga movement intervention (Active Comparator): Pre-recorded video of yoga movement intervention (Les Mills BodyBalance: mixture of yoga, tai chi, pilates) two times per week
  Interventions: Behavioral: Yoga movement intervention
- Education (Active Comparator): Education control group using a recently published postpartum physical activity guidebook through the Sport Information Resource Center
  Interventions: Other: Education booklet

INTERVENTIONS:
Behavioral: Yoga movement intervention — Mixture of yoga, tai chi, pilates. Will be delivered in person (experimental) and online (active comparator)
  Other Names: Les Mills BodyBalance; Les Mills BodyFlow
  Arms: In person movement intervention; Online yoga movement intervention
Other: Education booklet — Recently published postpartum physical activity guidebook through the Sport Information Resource Center of Canada
  Arms: Education

SUMMARY:
This is a mixed-methods randomized controlled trial assessing the effects of an online and in person 12-week movement intervention compared to an education only control group on heart rate variability, self-compassion, psychological well-being, fatigue, exercise self-efficacy, physical activity identity, and body image in postpartum women.

DETAILED DESCRIPTION:
This is a mixed-methods randomized controlled trial assessing the effects of an online and in person 12-week movement intervention compared to an education only control group on heart rate variability, self-compassion, psychological well-being, fatigue, exercise self-efficacy, physical activity identity, and body image in postpartum women.

Participants will be randomized into one of three groups: 1) in person yoga movement intervention, 2) online yoga movement intervention, 3) education group. Heart rate variability will be measured using a chest strap at the beginning and end of the 12 week intervention. At the beginning and end of the 12 week intervention, and at 3-months post-intervention, questionnaires will be completed online to assess self-compassion, psychological well-being, fatigue, exercise self-efficacy, physical activity identity, and body image.

ELIGIBILITY:
Inclusion Criteria:

* Women who have given birth to a child within the past 6 months and who are cleared for physical activity by their health care provider.

Exclusion Criteria:

* Participants who have a medical condition that precludes them passing the Get Active questionnaire
* Women not clear for physical activity by a health care provider
* Participants who are not able to attend classes at pre-specified times

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | Baseline, 12 weeks
  Waking RMSDD heart rate variability (chest strap)
Self compassion | Baseline, 12 weeks, 3 months
  Self-compassion scale, maximum score 125. Minimum score 25. Higher score is a better outcome.

SECONDARY OUTCOMES:
Physical activity | Baseline, 12 weeks, 3 months
  Type, amount and frequency of planned exercise, and walking bouts
Self efficacy | Baseline, 12 weeks, 3 months
  Self-efficacy and barrier to exercise scale. Maximum score of 36. Minimum score of 9. Lower score is a better outcome.
Fear of self-compassion | Baseline, 12 weeks, 3 months
  Fear of self-compassion scale. Maximum score of 60. Minimum score of 0. Lower score is a better outcome.
Fatigue | Baseline, 12 weeks, 3 months
  Multidimensional fatigue inventory scale. Maximum score is 100. Minimum score is 20. Lower score is a better outcome.
Sleep quality | Baseline, 12 weeks, 3 months
  Patient Reported Outcomes Measurement Information System (PROMIS) sleep questionnaire. Maximum score of 40. Minimum score of 8. Lower score is a better outcome.
Perceived stress | Baseline, 12 weeks, 3 months
  Perceived stress scale. Maximum score of 40. Minimum score of 0. Lower score is a better outcome.
Physical activity identify | Baseline, 12 weeks, 3 months
  Athlete identity measurement scale. Maximum score of 49. Minimum score is 7. Higher score is better outcome.
Body image | Baseline, 12 weeks, 3 months
  Body dissatisfaction scale. Maximum score of 48. Minimum score of 8. Lower score is better outcome.
Motivation for exercise | Baseline, 12 weeks, 3 months
  Psychological needs for exercise scale. Maximum score of 55. Minimum score of 11. Higher score is better outcome.
Postpartum depression | Baseline, 12 weeks, 3 months
  Edinburgh postnatal depression scale. Maximum score is 30. Minimum score is 0. Lower score is better outcome.
Anxiety | Baseline, 12 weeks, 3 months
  State-trait anxiety scale. Maximum score of 80. Minimum score of 20. Higher score is better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Lesser, PhD, Principal Investigator — University of the Fraser Valley; Gillian Hatfield, PhD, Principal Investigator — University of the Fraser Valley; Amanda Wurz, PhD, Principal Investigator — University of the Fraser Valley
Locations (1):
- University of the Fraser Valley, Chilliwack, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No